CLINICAL TRIAL: NCT06470230
Title: RESPECT: (REsearching Stigma in PEdiatric Cancer Tool)
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RESPECT; P30CA021765-44S2 (NIH)
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Stigma
Keywords: Cancer Related Stigma; Pediatric Cancer Population; Parent/Caregivers; Patients/Survivors; Diverse global settings
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric oncology patients/survivors: Children who have or had cancer
- Guardians/caregivers of pediatric oncology patients/survivors: Parents or caregivers of children who have or had cancer

SUMMARY:
Researchers want to learn more about the way stigma affects children with cancer and their caregivers. They want to develop two clinical tools to identify and measure stigma in the pediatric cancer population within culturally diverse global settings of the United States, Guatemala, and Jordan.

Primary Objectives

* Develop two clinical tools that can be used to identify and measure stigma as experienced by (1) pediatric oncology patients/survivors and (2) their guardians/caregivers in culturally diverse global settings.
* Pilot new stigma tools in geographically and culturally diverse cancer referral settings in the United States, Guatemala, and Jordan.

DETAILED DESCRIPTION:
There are 2 parts to this study; participants will be included in either Part 1 or Part 2, but not both.

In Part 1 of the study, investigators will conduct a systematic literature review of tools measuring stigma in healthcare at the level of the patient and survivor, or caregiver, through which they will catalog all items included in existing instruments of the study. Literature will be searched for concepts of patient self-stigma and scales, instruments, measurements, or outcomes.

Once the search strategy is completed, a panel of experts will review items and domains sorts to remove confusing or duplicative items and produce final pilot tools containing patient-centered and clinically relevant items. Preliminary tools will be translated into Spanish and Arabic. The preliminary English tools will be professionally translated into Spanish and Arabic. Translated tools will be reviewed by international study teams as well as bilingual members of the St. Jude team to account for regional linguistic differences. The Spanish and Arabic tools will be back translated into English to ensure original intent is maintained. Any modifications needed to ensure language consistency across versions will be made in all languages, ensuring parallel versions of the tool are developed.

We will recruit up to 20 active patients and/or survivor participants aged 8-17.9 in each language (up to 60 total patient/survivor participants), and similar numbers of parents or caregivers (not recruited as dyads) and ask questions about stigma. Experienced interviewers trained by the St. Jude team will verbally administer the tool followed by probing questions to assess face validity and rate each item on a scale of 1-5 based on accuracy, clarity, and difficulty of content. After 3-4 participants have been interviewed in each language, all three tools will be reassessed with modifications made as necessary. This process will be repeated until no additional modifications are identified through interviews.

In Part 2 of the study, children who have or had cancer and their caregivers will test out the questionnaire that was created during Part 1 of the study. Investigators will recruit 225-600 active patients or survivor participants (75-200 in each language) and 225-600 parents or caregivers (75-200 in each language) to pilot the tools.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive Debriefing and Pilot Data Collection - Patients/Survivors

  * Age 8 to 17.9 years of age
  * Active cancer patients or survivors of cancer
* Cognitive Debriefing and Pilot Data Collection - Parent/Caregivers

  * Adult parents or caregivers (≥ 18 years of age) of active cancer patients or survivors of cancer.

Exclusion Criteria: NA

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Active cancer patients or survivors of cancer and adult parents or caregivers of active cancer patients or survivors of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1320 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Develop two clinical tools that can be used to identify and measure stigma as experienced by (1) pediatric oncology patients/survivors and (2) their guardians/caregivers in culturally diverse global settings. | Up to 2 months after the start of study
  Concept mapping, a mixed-methods approach, combining qualitative group brainstorming and sorting with descriptive statistical analysis will be utilized to describe ideas and represent them graphically. Content expert participants, including members of the research team and global healthcare professionals, will generate novel items by answering prompts. Participants will sort the items into distinctive themes and conduct cluster analyses to create an initial concept map that improves understanding of stigma domains and will be asked to rate the importance and feasibility of each item. A panel of experts will review the item and domain sorts and ratings to remove confusing or duplicative items and produce final pilot tools containing patient-centered and clinically relevant items. Pragmatic design principles will be used to make the tools short and easy to use in a variety of settings.
Pilot new stigma tools in geographically and culturally diverse cancer referral settings. | Approximately one year after the start of study
  Pilot data will be analyzed using R. Data will be descriptively analyzed before psychometric analysis focusing on item- and domain-level characteristics, including inter-item correlation and scale internal consistency (Cronbach's alpha). Confirmatory factor analysis will test the structural validity (i.e., dimensionality) of the tools. The tools will be refined by dropping items, changing domains, or editing language. The analyses will highlight items that have poor fit and the expert team will review these items and make relevant updates to the overall measure based on these analyses and feedback regarding usability. This will result in a final version of the tools in all three languages.

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Graetz, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (4):
- United States (2):
  - Washington University School of Public Health, St Louis, Missouri
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- UNOP Unidad Nacional De Oncologia Pediatrica, Guatemala City, Guatemala
- King Hussein Cancer Center, Amman, Jordan

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols